CLINICAL TRIAL: NCT03491293
Title: Piloting Visual Chat in Internet Obesity Treatment
Acronym: CHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of South Carolina (Other); University of Tennessee (Other)
Responsible Party: Principal Investigator, Jean R. Harvey, PhD, RD, Principal Investigator, NFS Chair, Associate Dean, College of Agriculture and Life Sciences, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-0409
Record Dates: First submitted 2018-03-22; First posted 2018-04-09 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Obesity
Keywords: internet; behavioral weight loss; obesity
MeSH Terms: conditions — Obesity | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Weight Loss + Text chat (Active Comparator): Internet delivery of a behavioral weight control program via text in a group format facilitated by an experienced registered dietitian. Participants will have access to study materials including behavioral weight loss lessons on the study's website. Participants will weigh themselves daily and report their weight privately (data will only be accessible by research personnel) on the study website.
  Interventions: Behavioral: Behavioral Weight Loss + Text
- Behavioral Weight Loss + Video chat (Experimental): Internet delivery of a behavioral weight control program via video in a group format facilitated by an experienced registered dietitian. Participants will have access to study materials including behavioral weight loss lessons on the study's website. Participants will be given smart scales to weigh daily, and weight will be transmitted to a secure website accessible only by research personnel.
  Interventions: Behavioral: Behavioral Weight Loss + Video

INTERVENTIONS:
Behavioral: Behavioral Weight Loss + Text — Participants will attend weekly one hour classes on line. They will type their input and responses within the chat room. They will record their calorie and fat intake daily and weigh themselves daily. Interventionists will review the diaries weekly and provide feedback to reinforce or shape new behaviors and to identify high risk situations for problem solving.
  Arms: Behavioral Weight Loss + Text chat
Behavioral: Behavioral Weight Loss + Video — Participants will attend weekly one hour classes on line. They will have audio and video within the chat room, and will talk with their facilitator and classmates during their weekly meeting. They will record their calorie and fat intake daily and weigh themselves daily. Interventionists will review the diaries weekly and provide
  Arms: Behavioral Weight Loss + Video chat

SUMMARY:
CHAT is an internet-based weight loss research program designed for women with overweight or obesity who want to lose weight through dietary change and increased physical activity. Participants will be randomized into a group-based online program who meet via a text chat or a video chat.

DETAILED DESCRIPTION:
The overall goal of this project is to determine whether weight losses can be improved if visual chat and electronic smart scales are added to an established 6-month online weight loss program. The primary aim is to assess weight change differences between subjects randomized to receive an Internet program alone (with text chat; INTERNET) vs. an Internet program with visual chat and electronic scales (VIDEO INTERNET). A secondary aim is to evaluate differences in social support experienced by subjects in both conditions. Overweight and obese adults (n=40) at two study sites (UVM and the University of South Carolina) will be randomly assigned to Internet (n=20) or Video Internet (n=20). All participants will receive the same 24 week web-based group weight control program which features synchronous facilitated chats and online behavioral tools. The only difference will be the delivery of the chat (text vs. visual) and the electronic smart scales given to the VIDEO INTERNET group. Assessments will be conducted at 0, 2 and 6 months and will include measures of body weight, treatment engagement (e.g., attendance, self-monitoring, website utilization), social support and treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* BMI between 25 and 55
* Free of medical problems that would preclude participation in a behavioral weight reduction program containing an exercise component
* Not currently pregnant or pregnant in the previous 6 months or breastfeeding
* Must have a computer at home or work with access to the Internet
* Only one member of a household is eligible to participate
* Must successfully complete a self-monitoring diary of foods consumed for 3 days
* must be willing to share access to self monitoring information collected via My Fitness Pal by friending the CHAT research team
* Not currently on medication that might affect weight loss
* Not enrolled in another weight loss program

Exclusion Criteria:

* BMI less than 25 or more than 55
* Lost 10 pounds or more in the last 6 months
* Had a heart attack or stroke in the past 6 months
* Ever had weight loss surgery
* Currently taking medications for weight loss
* Persons required by their doctor to follow a special diet (other than low fat)
* Plans to move from the area in the upcoming 9 months
* Schedules that make it likely someone would have difficulty attending the scheduled chat groups

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Weight loss from baseline | baseline, 2 months, 6 months
  The investigators will assess weight change differences between subjects randomized to receive an internet program alone with text chat vs. an internet program with visual chat and bodytrace smart scales. Weight will be assessed at baseline, 2 months after intervention begins, and at the end of intervention using a calibrated digital scale (Tanita, WB800S) with subjects in street clothes, without shoes.

SECONDARY OUTCOMES:
Attendance at chat | 6 months
  The group facilitator will record attendance at chats. Attendance at chat will be compared by treatment arm. Rate of attendance is calculated as number of meetings attended out of a total possible 24 meetings over the course of the study.
Self monitoring dietary intake | 6 months
  Number of weekly journals submitted out of a possible 24 weeks total will give the investigators the rate of self monitoring. Rates of self monitoring will be compared by treatment arm.
Self monitoring weight | 6 months
  Number of daily weights submitted over the course of 24 weeks divided by the possible total of weights will give the rate of weight self-monitoring (7/week x 24 weeks = 168 possible weights). The VIDEO arm will be provided with BodyTrace electronic scales that report weight to a secure database via cellular connectivity. Subjects in the TEXT arm will report their weights to their facilitator using their own digital scale at home.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Harvey, PhD RDN, Principal Investigator — University of Vermont; Delia West, PhD, Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - University of South Carolina, Columbia, South Carolina
  - Behavioral Weight Management Program/Univ of Vermont, Burlington, Vermont